CLINICAL TRIAL: NCT05480358
Title: Phase I/II Randomized Clinical Trial of a Low Protein Diet in Patients With Cognitive Impairment
Brief Title: Clinical Trial of a Low Protein Diet in Patients With Cognitive Impairment
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Genova (Other)
Responsible Party: Principal Investigator, Alessio Nencioni, Full Professor, University of Genova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMD AD
Record Dates: First submitted 2021-10-18; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Mild Cognitive Impairment; Mild Dementia; Fasting-Mimicking Diet
Keywords: Fasting-Mimicking Diet; nutritional status; MCI; Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: This is a pilot, double arm randomized and prospective clinical trial assessing feasibility and safety of a 5-day low protein fasting-mimicking diet in pazients affected by Mild Cognitive Impairment or early Alzheimer disease.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ProlonADTM (Experimental): The ProlonADTM diet, which will be taken by the patient once a month for 5 days, is a low-calorie and low-protein diet, and provides all the micronutrients necessary to avoid malnutrition. The diet will be performed in twelve consecutive months. The components of the diet will be approximately 30% calorie restricted and 50% protein restricted but supplemented with 50% of the RDA in vitamins and minerals and also supplemented with both nonessential and essential amino acids identified in animal studies to be effective. Prolon by L-Nutra is a medically-designed dietary kit providing the food to eat for five days. Day 1 of Prolon provides ~4600 kJ (11% protein, 46% fat, and 43%carbohydrate), whereas days 2-to-5 provide ~3000 kJ (9% protein, 44% fat, and 47% carbohydrate) per day.
  Interventions: Dietary Supplement: Fasting-Mimicking Diet ProlonADTM
- Placebo diet (Placebo Comparator): One meal which substitute or lunch or dinner for 5 days, without calories restriction.
  Interventions: Dietary Supplement: Fasting-Mimicking Diet ProlonADTM

INTERVENTIONS:
Dietary Supplement: Fasting-Mimicking Diet ProlonADTM — Prolon by L-Nutra is a medically-designed dietary kit providing the food to eat for five days. Day 1 of Prolon provides ~4600 kJ (11% protein, 46% fat, and 43% carbohydrate), whereas days 2-to-5 provide ~3000 kJ (9% protein, 44% fat, and 47% carbohydrate) per day.

SUMMARY:
The wide-acting effects of Fasting-Mimicking Diets (FMDs) on metabolic, inflammatory and regenerative pathways leading to reduced pathology or risk factors for various diseases in mice and humans, has the potential to be effective against Alzheimer's disease (AD). It is proposed to conduct a randomized clinical trial of twelve monthly cycles of the ProlonADTM diet (by L-Nutra) vs. placebo diet in patients with aMCI or mild AD (MMSE 18-23). The primary endpoint of the study will be the feasibility and safety of the twelve cycles of ProlonADTM.

DETAILED DESCRIPTION:
Cognitive impairment that exceeds the physiological decline associated with aging can take the form of mild cognitive impairment (MCI) or, in its most severe form, dementia. In turn, patients diagnosed with MCI evolve towards outright Alzheimer's disease (AD) in an estimated percentage of 15%/year. MCI can occur in the form of amnestic MCI (amnestic MCI, aMCI; by far the most common) or non-amnestic MCI (single or multiple domain), where amnestic is the form that most frequently evolves into AD. Therefore this clinical trial will focus on the latter (as well as on the AD). Diet cycles with low sugar and protein levels followed by diets with normal levels of these lead to temporary reductions in growth hormone and IGF-1 levels. Both are potential mediators of the neuroprotective and regenerative effects of these diets not only in mice, but also in monkeys and humans . However, heavily restricted diets in terms of calories are often difficult to endure over time and are frequently associated with side effects, even significant ones and with progressive weight loss, in particular of lean mass. In a mouse model of AD, it has been shown that periodic cycles of a "fasting-mimicking" diet (FMD) restricted in protein content (PR-FMD) but not in terms of calories are able to reduce levels plasma levels of IGF-1 with contrasting effects on the neurodegeneration process. In particular, such FMD has been shown to reduce by about 30-70%, the levels of hyperphosphorylated tau protein (one of the typical markers of AD) at the hippocampal level, reducing the age-related deficit of cognitive performance. A relevant neuroregenerative effect (associated with a clinical improvement in motor coordination and memory) has been demonstrated in mice subjected to a diet based on a similar DMD during their "average life" (months 16-30).

It is proposed to conduct a study of twelve monthly cycles of the ProlonADTM diet (by L-Nutra) in patients with aMCI or mild AD (MMSE 18-23) diagnosed according to the criteria defined by Peterson and McKahn, respectively (1, 3 ).

It is proposed to conduct a randomized clinical trial of twelve monthly cycles of the ProlonADTM diet (by L-Nutra) vs. placebo diet in patients with aMCI or mild AD (MMSE 18-23). Patients in the treatment group alone will also receive a range of supplements containing omega-3 fatty acids, caffeine, tree nuts, coconut oil, olive oil and cocoa - which will be supplied with the ProlonADTM diet kit. Patients assigned to both arms will also receive personalized dietary recommendations matched to instructions for light-moderate physical activity to be carried out also at home and aimed, especially in the case of patients assigned to receive ProlonADTM, to prevent the loss of lean mass. The primary endpoint of the study will be the feasibility and safety of the twelve cycles of ProlonADTM. Feasibility is defined as taking at least one course of DMD every two months with the option of admitting consumption of 50% of the planned diet and / or a maximum consumption of 10 Kcal / kg of unforeseen food in only one of days 1-5 of each cycle. Investigators speculate that ProlonADTM will not cause severe side effects and that it will have no detrimental effect on the patient's body composition, specifically in terms of impact on lean mass measured by dynamometry and bioimpedance analysis.

Secondary objectives will include:

* conversion rate to AD (for patients with aMCI);
* episodic memory evaluated with Free and Cued Selective Reminding Test (FCRST);
* cognitive status assessed by MMSE, CDR-Sum of the boxes;
* functional status assessed with Barthel Index, IADL;
* emotional state assessed using the CESD-R scale;
* nutritional status (MNA and body composition - bioimpedance, handgrip);
* caregiver stress assessed through Caregiver Burden Inventory and NPI;
* quality of life of patients (QLQ-AD);
* inflammatory markers, oxidative stress markers, neuronal damage markers (Neurofilament Light, NfL), quantification of circulating stem cells, cell aging markers (eg evaluation of the telomerase activity of lymphocytes).
* assessment of frailty (Rockwood frailty index, which also includes walking speed, handgrip, breathing capacity)

ELIGIBILITY:
Inclusion Criteria:

* Age 55-80;
* Presence of aMCI or initial AD (MMSE 18-23);
* Normal organ function (liver and kidney);
* BMI not less than 20 kg/m2;
* Bioimpedance phase angle (PA) > 5 °;
* Adherence to informed consent

Exclusion Criteria:

* Age> 80 years
* Diabetes mellitus;
* Organ impairment (liver, kidney);
* Food allergies to the components of ProlonADTM;
* Patients on therapy with vitamin K antagonist anticoagulants;
* PA <5 °;
* Patients who live alone or are not adequately supported by the family context;
* Other experimental therapies in progress.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 12 months
  Safety of FMD in terms of percentage of patients experiencing adverse events and/or worsening of nutritional status.
  To obtain clinical data on safety of the FMD in MCI or AD patients as assessed by percentage of patients (%) experiencing > grade 3 adverse events and/or a significant decrease in their lean body mass (kg) and/or with a reduction of phase angle <5° assessed with bio-impedance measurements.
Percentage of patients able to achieve the designated diet regimen | 12 months
  Feasibility of FMD in terms of percentage of patients able to complete the diet regimen To evaluate the feasibility of the FMD in MCI and AD patients as assessed by the percentage of patients (%) able to achieve the designated diet regimen.

SECONDARY OUTCOMES:
Efficacy of the FMD in terms of conversion rate to AD | 12 months
  Efficacy of the FMD in terms of coversion rate to AD will be assessed with the conversion rate (%) from AD to aMCI
Efficacy of the FMD in terms of functional state | 12 months
  Efficacy of the FMD in terms of functional will be assessed with Barthel Index (BI) from 0 as the worse score and 100 as the best score.
Efficacy of the FMD in terms of emotional state | 12 months
  Efficacy of the FMD in terms of emotional state will be assessed with the Center for Epidemiologic Studies Depression Scale Revised (CESD-R) with 0 as the best score and 80 as the worse score.
Efficacy of the FMD in terms of nutritional state | 12 months
  Efficacy of the FMD in terms of nutritional state will be assessed with phase angle with bioimpedance (°)
Efficacy of the FMD in terms of caregiver stress' level | 12 months
  Caregiver stress will assessed through Caregiver Burden Inventory (CBI) with 0 as the best score and 96 as the worse score
Efficacy of the FMD in terms of quality of life | 12 months
  Efficacy of the FMD in terms of quality of life of patients with Quality of Life AD (QLQ-AD) with 13 as the worse score and 52 as the best score.
Efficacy of the FMD in terms of prevention of Frailty | 12 months
  Efficacy of the FMD in terms of prevention of Frailty with 40-item Rockwood frailty index (FI) with 0 as the best score and 1 as the worse score.
Efficacy of the FMD in terms of alzheimer and inflammatory biomarkers | 12 months
  We will assess the inflammatory markers, oxidative stress markers, neuronal damage markers (Neurofilament Light, NfL), quantification of circulating stem cells, cell aging markers (eg evaluation of the telomerase activity of lymphocytes)
Efficacy of the FMD in terms of episodic memory | 12 months
  Efficacy of the FMD in terms of episodic memory will evaluated with Free and Cued Selective Reminding Test (FCRST) with a range from 0 as worse score to 36 as best score.
Efficacy of the FMD in terms of general cognitive status | 12 months
  Efficacy of the FMD in terms of general cognitive status with mini-mental state examination (MMSE) with 0 as worse score and 30 as the best score.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Alessio Nencioni, Genoa, GE
  - Ospedale Policlinico San Martino, Genova
  - Azienda Ospedaliera di Perugia, Perugia

REFERENCES:
- [Derived] Rangan P, Lobo F, Parrella E, Rochette N, Morselli M, Stephen TL, Cremonini AL, Tagliafico L, Persia A, Caffa I, Monacelli F, Odetti P, Bonfiglio T, Nencioni A, Pigliautile M, Boccardi V, Mecocci P, Pike CJ, Cohen P, LaDu MJ, Pellegrini M, Xia K, Tran K, Ann B, Chowdhury D, Longo VD. Fasting-mimicking diet cycles reduce neuroinflammation to attenuate cognitive decline in Alzheimer's models. Cell Rep. 2022 Sep 27;40(13):111417. doi: 10.1016/j.celrep.2022.111417. PMID 36170815